CLINICAL TRIAL: NCT00420407
Title: Prospective, Randomized, Double-Blind, Multi-Center Trial of Low Dose Vasopressin Versus Placebo in Traumatic Shock Resuscitation
Brief Title: Low Dose Vasopressin in Traumatic Shock
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: accrual rate
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 056-1502-090
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2013-04

CONDITIONS: Injuries; Shock, Traumatic
MeSH Terms: conditions — Wounds and Injuries; Shock, Traumatic | interventions — Vasopressins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- I (Experimental): Vasopressin
  Interventions: Drug: vasopressin
- 2 (Placebo Comparator): bolus of NS (normal saline) followed by continuous infusion of NS, no vasopressin added
  Interventions: Drug: normal saline control

INTERVENTIONS:
Drug: normal saline control — no vasopressin added to bolus or 5 hour continuous infusion
  Arms: 2
Drug: vasopressin — vasopressin bolus 4 units followed by continuous infusion 2.4units/hr for 5 hours
  Arms: I

SUMMARY:
Hypothesis: We hypothesize that resuscitation regimens which minimize the total volume of resuscitation fluid, while restoring organ perfusion, will lead to lower morbidity and mortality in critically ill patients following trauma.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment in the study, a patient must meet all of the follow criteria at assessment:

* Patient is a male or female patient presumed to be at least 18 years of age;
* Patient has a systolic blood pressure < 90 mmHg;
* Patient has clinical evidence of acute traumatic injury;
* Infusion of study drug must start within one hour following SBP (systolic blood pressure) < 90 mmHg

Exclusion Criteria:

A patient meeting any one of the following criteria at hospital assessment is not eligible for enrollment:

* Patient is admitted to one of the study hospitals' Emergency Department greater than six hours after injury;
* Patient has received greater than 4 liters fluid since time of injury;
* Patient is enrolled in another shock trial;
* Patient is asystolic or requires CPR (cardiopulmonary resucitation) prior to randomization;
* Female patient is pregnant by report or suspicion;
* Patient has known "Do Not Resuscitate" orders or visible/identifiable method of objection to participation (e.g., exclusion bracelet);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M. Cohn, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Result] Cohn SM, McCarthy J, Stewart RM, Jonas RB, Dent DL, Michalek JE. Impact of low-dose vasopressin on trauma outcome: prospective randomized study. World J Surg. 2011 Feb;35(2):430-9. doi: 10.1007/s00268-010-0875-8. PMID 21161222
- See also: Department of Surgery Web Page, Vasopressin presentation — http://www.surgery.uthscsa.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment location - Emergency room Feb 2007- Feb 2009
Pre-assignment Details: clinical indication prohibiting potential use of vasopressin.
Groups:
- Normal Saline: bolus of NS (normal saline) followed by continuous infusion of NS, no vasopressin added
  normal saline control : no vasopressin added to bolus or 5 hour continuous infusion
- Vasopressin: Vasopressin
  vasopressin : vasopressin bolus 4 units followed by continuous infusion 2.4units/hr for 5 hours
Period: Overall Study
Arm/Group | Normal Saline | Vasopressin
Started | 41 | 40
Completed | 37 | 34
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 0 | 3
Not completed — Physician Decision | 2 | 1
Not completed — subject identified as detainee | 1 | 0
Not completed — subject identified as Jehovah's witness | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Vasopressin enrolled 40 and two withdrawn and never received drug (38) Normal saline enrolled 41 and one withdrawn and never received drug (40)
Groups:
- Normal Saline: bolus of NS followed by continuous infusion of NS, no vasopressin added
  normal saline control : no vasopressin added to bolus or 5 hour continuous infusion
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Vasopressin | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (26.1) | 48.1 (19.8) | 47.1 (20.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 34 | 29 | 63
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Study Will be Day 30 Mortality.
Description: Survival of a traumatic injury subject to at least 30 days after admission to the emergency room.
Time Frame: 30 days
Measure: Number; unit: Participants
Groups:
- Vasopressin: vasopressin : vasopressin bolus 4 units followed by continuous infusion 2.4units/hr for 5 hours
Arm/Group | Normal Saline | Vasopressin
Number analyzed (Participants) | 37 | 34
Participants | 11 | 13

2. Secondary Outcome: Level of Vasopressin After Trauma.
Description: Level of vasopressin 12 hours after infusion was measured for all subjects in vasopressin arm
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Evaluation of Vasopressin Level Following Trauma: All traumatic subjects that had a blood sample assessed for vasopressin.
Arm/Group | Evaluation of Vasopressin Level Following Trauma
Number analyzed (Participants) | 34
pg/ml | 25 (37)

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after Day 0 or before Day 30
Arm/Group | Normal Saline | Vasopressin
Serious Adverse Events (participants affected / at risk) | 19/41 | 20/40
Other Adverse Events (participants affected / at risk) | 37/41 | 35/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=41) | Vasopressin (N=40)
Cardiopulmonary Arrest (General disorders) | 4 (4) | 3 (3) — includes cardiac and cardiopulmonay arrest
Cardiac Dysrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
exsanguination (General disorders) | 1 (1) | 1 (1)
Hemorrhagic Shock (General disorders) | 1 (1) | 3 (3) — includes refractory hemorrhagic shock(1)
Hypertenson (Cardiac disorders) | 0 (0) | 2 (2)
Multisystem Trauma (General disorders) | 3 (3) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2) — Pulseless electrical activity, pulseless ventricular tachycardia, supraventricular tachycardia, intermittent
reperfusion syndrome (Vascular disorders) | 0 (0) | 1 (1)
Ogilvies Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper GI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 3 (3) — locations - Femoral, popliteal, subclavian
Heparin induced thrombocytopenia (Vascular disorders) | 0 (0) | 1 (1)
Sepsis, abdominal (General disorders) | 0 (0) | 1 (1)
Dehiscence, wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Systemic Inflamatory Response Syndrome (SIRS) (General disorders) | 1 (1) | 0 (0)
Ischemic Necrosis Bilateral Lower Extremities (Vascular disorders) | 0 (0) | 1 (1)
Bacterial Meningitis (General disorders) | 1 (1) | 0 (0)
Cellutlitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Shock, Septic (General disorders) | 1 (1) | 0 (0)
Multiple Organ Failure (General disorders) | 2 (2) | 4 (4) — includes multiple organ dysfunction.
Compartment Syndrome (Vascular disorders) | 0 (0) | 1 (1)
Traumatic Brain Injury (TBI) (Nervous system disorders) | 3 (3) | 4 (4) — nonsurvivable TBI
Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Empyema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pulmonary Emboli (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) — included pulmonary embolis and embolism
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Retroperitoneal bleed (General disorders) | 1 (1) | 0 (0)
Pulmonary Hemorrhage (General disorders) | 0 (0) | 1 (1)
Renal Insufficiency, worsening (Renal and urinary disorders) | 0 (0) | 1 (1)
Candidemia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=41) | Vasopressin (N=40)
Hypotension (Cardiac disorders) | 2 (2) | 3 (3)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Hypoperfusion (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Adrenal Insufficiency (Endocrine disorders) | 4 (4) | 0 (0)
Diabetes Insipidus (Endocrine disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 9 (9) | 6 (6) — included intermittent Hyperglycemia
hypoglycemia (Endocrine disorders) | 1 (1) | 2 (2) — includes intermittent hypoglycemia
Hyperphosphatemia (Endocrine disorders) | 1 (1) | 0 (0)
Hypocalcemia (Endocrine disorders) | 5 (5) | 3 (3) — includes intermittent hypocalcemia
Hypokalemia (Endocrine disorders) | 5 (5) | 4 (4) — includes intermittent hypokalemia
Hypomagnesemia (Endocrine disorders) | 2 (2) | 1 (1) — included intermittent hypomagnesemia
Hypophosphatemia (Endocrine disorders) | 7 (7) | 2 (2) — includes intermittent hypophosphatemia
Dysphagia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Thrush (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypernatremia (Endocrine disorders) | 1 (1) | 0 (0) — includes intermittent hypernatremia
Hyponatremia (Endocrine disorders) | 1 (1) | 0 (0) — includes intermittent hyponatermia
Hyperkalemia (Endocrine disorders) | 0 (0) | 1 (1) — includes intermittent hyperkalemia
Otorrhea (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Acute Choleycystitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bowel Distention (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 5 (5) — includeds intermittent
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Elevated gastric residuals (Gastrointestinal disorders) | 1 (1) | 2 (2)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
incontinence stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) — includes intermittent
oliguria (Renal and urinary disorders) | 2 (2) | 0 (0) — Urinary retention, failur to void
Incontinence Urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 4 (4) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Dilitional Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Elevated INR (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cephalic Vein Thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Elevated Liver Function Tests (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal Infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 2 (2) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Elevated Temperature (Infections and infestations) | 2 (2) | 2 (2)
Postitive blood cultures (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 3 (3) | 2 (2)
Skin Breakdown (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (8)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infiltration, skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Itching, intermittant (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Multiorgan failure (General disorders) | 6 (6) | 3 (3) — Hepatic/pulmonary
Rhabdomyolosis (General disorders) | 1 (1) | 0 (0)
Myoglobinuria (General disorders) | 0 (0) | 1 (1)
Edema (Vascular disorders) | 0 (0) | 1 (1) — bilateral lower extremity edema
Agitation (Nervous system disorders) | 1 (1) | 1 (1)
Allergic reaction to enalapril (General disorders) | 1 (1) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Delirium Tremors (Nervous system disorders) | 1 (1) | 1 (1)
Azotemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Elevated Lactic Acid (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hiccups (General disorders) | 1 (1) | 0 (0)
Hyper-reflexia (Nervous system disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 2 (2) | 1 (1) — included intermittent
insomia (Nervous system disorders) | 5 (5) | 1 (1) — included intermittent
anxiousness (Nervous system disorders) | 1 (1) | 0 (0) — intermittent
Hyperchloremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — intermittent
Pain (General disorders) | 1 (1) | 2 (2)
Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Impaired Renal Function (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) — unilateral and/or bilateral
Exacerbation COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — intermittent
Laryngeal Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — includes lung infection
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No